CLINICAL TRIAL: NCT01719107
Title: Efficacy of Dietary Supplementation With Lactobacilllus Reuteri DSM 17938 on Functional Abdominal Pain (FAP) in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aghia Sophia Children's Hospital of Athens (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Alexandra Papadopoulou, Consultant in Pediatrics, Honorary Professor Dr. med., Aghia Sophia Children's Hospital of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUB0003
Record Dates: First submitted 2012-10-28; First posted 2012-11-01 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Functional Abdominal Pain (FAP) in Children
Keywords: Functional abdominal pain; Probiotics; Lactobacilus reuteri

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L. reuteri DSM 17938 chewable tablets (Active Comparator): The active study product consists of a citrus flavored 450 mg chewable tablet containing freeze-dried L. reuteri DSM 17938. The study product is a convex tablet 10.3 mm in diameter, plain on both sides and with faint spots. It is composed of freeze-dried L. reuteri, isomalt, xylitol, sucrose distearate, hydrogenated palm oil, lemon-lime flavoring and anhydrous citric acid. The total viable count of L. reuteri DSM 17938 is 1x108 live bacteria (CFU)/tablet.
  Interventions: Dietary Supplement: L. reuteri DSM 17938 chewable tablets
- Placebo chewable tablets (Placebo Comparator): The placebo study product consists of an identical formulation in all respects except that the live bacteria are excluded.
  Interventions: Dietary Supplement: Placebo chewable tablets

INTERVENTIONS:
Dietary Supplement: L. reuteri DSM 17938 chewable tablets — 2 chewable tablets with breakfast for 4 weeks
  Arms: L. reuteri DSM 17938 chewable tablets
Dietary Supplement: Placebo chewable tablets — 2 chewable tablets with breakfast for 4 weeks
  Arms: Placebo chewable tablets

SUMMARY:
The aim of the study is to investigate the effect of L. reuteri DSM 17938 on pain frequency and severity in children of 5-16 years old and with diagnosis of FAP.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study. Subjects between of 5-16 years of age with FAP as defined in the Rome III criteria and with pain severity of at least 40 mm on a 100 mm VAS scale and pain frequency of at least 1 episode per week over the preceding 8 weeks will be recruited. In accordance to the specific Rome III criteria for inclusion, FAP is defined as a variable combination of chronic or recurrent gastrointestinal symptoms not explained by structural or biochemical abnormalities.

A study questionnaire to record pain and other gastrointestinal symptoms will be used.

One-hundred and six (106) Subjects will be randomized to receive either dietary supplementation with L. reuteri DSM 17938 (2 chewable tablets with breakfast), or the same number of comparable placebo tablets, for 4 weeks. Supplementation will be stopped after 4 weeks, and the subjects will be followed up for an additional 4 weeks. The subjects will complete a diary to record frequency and intensity of pain, use of medication, deviation from the usual diet, physical activities, and absence from school and other activities. Gastrointestinal symptoms are assessed by the GSRS (Gastrointestinal Symptom Rating Score).

Subjects/caregivers will be instructed to maintain the usual diet throughout the study, but not to consume other probiotics (foods or supplements) during the entire study period.

The symptoms diary will be completed daily by the parents and will report information on the frequency of pain episodes, location of pain, presence or absence of associated symptoms, need to take medication for pain and interference with normal activities. The intensity of the symptoms will be assessed by using the Wong-Baker Faces scale.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be recruited according to the following inclusion criteria:

* FAP (Functional Abdominal Pain) according to Rome III criteria for Child/Adolescent; 1 or more abdominal pain episodes per week over the past 8 weeks
* Informed consent by study participant and at least one parent/legal guardian;
* Age of 5-16 years;
* Pain severity at study entry must be at least 40 mm on a 100 mm VAS scale;
* Pain frequency of at least 1 or more episodes per week over the preceding 8 weeks;
* Ability to understand and comply with the requirements of the trial;
* Stated availability throughout the study period

Exclusion Criteria:

Subjects presenting with one or more of the following criteria will be excluded from participation in the study:

* Chronic illness;
* Surgery of gastrointestinal tract
* Any symptoms/signs of organic disease and/or any abnormal results of laboratory assays (total blood count, serum glucose, urea, electrolytes, amylase, SGOT, SGPT, anti tTG antibodies, breath H2 test, suggesting disease other than FAP;
* Weight loss of 5% or more in body weight over the preceding 3 months;
* Exposure to any drugs for FAP in the past 2 weeks.
* Exposure to probiotics or antibiotics within 4 weeks prior to study; subjects can be included following a wash-out period of 4 weeks.
* Participation in other interventional clinical trials in the past 3 months;
* Subjects with special dietary needs

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Abdominal pain frequency and severity over the 4-week treatment period. | 4 weeks
  Reduction in pain frequency measured by a subject diary, in the L. reuteri DSM 17938 group and the placebo group, expressed as area under the pain-frequency curve and comparing L. reuteri DSM 17938 vs placebo over the treatment period.
  Reduction in pain severity is assessed using the face score system of Wong-Baker at day 14 and at the end of treatment (day 28)vs. baseline. Area under the pain-intensity curve will be assessed for Weeks 1-4 and Weeks 1-2

SECONDARY OUTCOMES:
Reduction in pain frequency and intensity over the 8-week study period | 8 weeks
  Reduction in pain frequency measured by a subject diary in the L. reuteri group expressed as area under the L. reuteri pain-frequency curve compared to placebo over the initial 2 weeks of the treatment period as well as over the whole study period.
  Reduction in pain intensity, measured by the face score system of Wong-Baker at day 14, end of treatment (day 28), and end of follow-up period (day 56) vs baseline. Area under the pain-intensity curve for Weeks 1-4 and Weeks 1-2 will be compared.
Reduction in other GI symptoms over the whole study period | 8 weeks
  Reduction in other GI symptoms as measured by Gastrointestinal Symptom Rating Scoring system. Time points: baseline, day 14, end of treatment and end of follow-up, in the L. reuteri group vs. placebo.
Days of absence from school and other activities due to abdominal pain over the whole study period | 8 weeks
  The number of days of absence from school and other activities due to abdominal pain will be compared between the L. reuteri group vs placebo.
Reduction in absence from work by parents over the whole study period | 8 weeks
  he number of days of absence from work by parents due to abdominal pain of the child will be compared between the L. reuteri group vs placebo.
Safety outcome over the whole study period | 8 weeks
  The number of adverse events will be observed and recorded during the entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papadopoulou, Hon. Prof. Dr. med., Principal Investigator — Athens Interconnected Children's Hospitals "AGIA SOPHIA" and "P & A KYRIAKOU"; Hania Szajewska, Prof, Principal Investigator — Warsaw University; Rok Orel, Ass. Prof., Principal Investigator — Ljubljana University
Locations (3):
- Athens Children's Hospital "AGIA SOPHIA", Athens, Attica, Greece
- University of Warsaw, Department of Pediatrics, Warsaw, Poland
- University of Ljubljana, Children's Hospital, Department of Gastroenterology, Ljubljana, Slovenia